CLINICAL TRIAL: NCT00225888
Title: Digital Photography and Group Discussion as a Means of Affecting Dietary Change Among People With Type 2 Diabetes: Feasibility Project
Brief Title: Feasibility Study of Digital Photography and Group Discussion for People With Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators left Joslin
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Stephanie Fonda, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS #03-47; DAMD17-03-2-0062
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Nutrition; Digital photography; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Snacks

INTERVENTIONS:
Behavioral: Digital Photography of meals/snacks and group discussion — Digital Photography of meals/snacks and group discussion

SUMMARY:
The purpose of this study is to compare the effect of food photography with group discussions to the effect of regular diabetes nutrition care on people's eating habits, satisfaction with care, self-care behaviors, and blood sugar levels. We hypothesize that, by photographing all meals and snacks (i.e., keeping 'photo journals') and participating in discussions about the photographs with peers and a nutritionist, people with diabetes will become aware of their behaviors and develop concrete strategies to meet nutritional recommendations.

DETAILED DESCRIPTION:
Diet is critical to effective self-management of diabetes. Thus, people with diabetes receive substantial nutrition counseling as part of their care. Among other things, nutrition counseling can include nutrition facts, information about portions, menus, discussion of barriers to healthy eating, and recommendations to control intake of saturated fats, maintain consistent eating patterns, and distribute nutrient intake throughout the day. Despite the depth and breadth of nutrition counseling, many people with diabetes implement diet changes with limited success.

The overall objective of this study is to test the feasibility of a new approach to diabetes nutrition care, digital food photography and facilitated group discussions. The overall hypothesis regarding this new approach is that, by photographing all meals and snacks (i.e., keeping 'photo journals') and participating in discussions about the photographs with peers and a nutritionist, people with diabetes will become aware of their behaviors and develop concrete strategies to meet nutritional recommendations. This overall hypothesis can be further specified as follows:

* People with diabetes who receive the new approach to diabetes nutrition care (i.e., the digital photos with discussions) will show greater improvements in their nutritional profiles and hemoglobin A1c (HbA1c) values (primary clinical outcomes) than people who receive standard diabetes nutrition care.
* People with diabetes who receive the new approach to diabetes nutrition care will become more satisfied with their diabetes treatment compared to people who receive standard care (secondary clinical outcome).
* People with diabetes who receive the new approach to diabetes nutrition care will show greater improvements in minimizing the barriers that affect their abilities for effective self-care compared to people who receive standard care (secondary outcome).

The study design is that of a single-site, randomized controlled trial with two groups of approximately 18 study participants assigned to each (for a total of 36 study participants). The study will take place at Joslin Diabetes Center. One group will receive standard diabetes nutrition care. The other group will receive the new approach to diabetes nutrition care involving digital photography of meals and group discussion of the photographs. All participants will complete study questionnaires before the study begins and approximately 1 month after the completion of the digital photography discussion groups.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient of the Joslin Diabetes Center
* Must have type 2 diabetes
* Must be between 30 and 60 years of age
* Must have a BMI equal to or greater than 30
* Must agree to randomization
* Must provide written informed consent

Exclusion Criteria:

* Unable to give written informed consent
* Unable to communicate in and read English
* A severe visual impairment
* Pregnancy
* Non-compliance or unlikely to return for the treatment

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-07-20 (Actual); Study Completion 2007-07-20 (Actual)

PRIMARY OUTCOMES:
Subjects' nutritional profiles | 6 months
Subjects' hemoglobin A1c (A1c) values | 6 months

SECONDARY OUTCOMES:
Subjects' satisfaction with diabetes treatment | 6 months
Subjects' self-care behaviors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J. Fonda, Ph.D., Principal Investigator — Joslin Diabetes Center and Harvard Medical School
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States